CLINICAL TRIAL: NCT00510731
Title: Prospective, Multi-Center Study Of The Ability Of The PD2i Cardiac Analyzer To Predict Risk Of VentrIcular TachyArrhythmic Events Such As, Sudden Cardiac Death, VentricuLar Fibrillation or Ventricular Tachycardia in High Risk Patients
Brief Title: The Ability Of The PD2i Cardiac Analyzer To Predict Risk Of Ventricular Tachyarrhythmic Events
Acronym: VITAL
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: Vicor Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VTI-2003-03
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Tachycardia, Ventricular; Cardiac Sudden Death
Keywords: Ventricular Tachycardia; Cardiac Sudden Death; Ventricular Fibrillation; Heart Rate Variability
MeSH Terms: conditions — Tachycardia, Ventricular; Death, Sudden, Cardiac; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a prospective study to evaluating the ability of the PD2i Cardiac Analyzer to predict the risk of serious heart rhythm abnormalities in high-risk patients that do not already have an Implantable Cardioverter Defibrillator.

DETAILED DESCRIPTION:
The annual incidence of sudden cardiac death in the United States has recently been estimated at 450,000. Most of these patients die from ventricular tachyarrhythmias. Currently, there is a limited ability to predict reliably which patients are at risk for these events. Implantable cardioverter defibrillators (ICDs) are highly effective at treating the arrhythmias that cause sudden death. Multiple clinical trials demonstrating the efficacy of ICDs for the primary prevention of sudden death have been completed, leading to a relaxation of the selection criteria for their use, and therefore a potentially large expansion in the pool of patients eligible for these devices. This has major economic implications for the health care system, and has led to a need for better prospective identification of patients who are or are not at high risk for sudden death.

The existence of beat-to-beat changes in heart rate, termed heart rate variability HRV), has long been recognized by physiologists. However, over the past 15 years, it has been determined that HRV is not a random phenomenon but can be influenced by the brain through the autonomic nervous system.

Promising work in the analysis of HRV may provide a means of predicting which patients are at risk for sudden death. HRV analysis utilizes mathematical modeling of ECG data to gain insight into the subtle variations in heartbeat patterns which occur from beat-to-beat.

The development of a system that could better identify the patients at risk of arrhythmic events would have a significant impact on clinical and economical fields. This study will test software developed by Vicor Technologies that can potentially identify patients at risk of arrhythmic events. It works as a generic digital-electrocardiogram (ECG) device, as it would normally be used by technical personnel in the routine care of outpatients.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Left Ventricular Ejection Fraction (LVEF) <35%
* Prior myocardial infarction
* Symptomatic congestive heart failure
* Referred for EP testing and/or prophylactic ICD implantation

Exclusion Criteria:

* Currently has implanted pacemaker or ICD
* Current atrial fibrillation/flutter or atrial fibrillation/flutter requiring cardioversion within the previous 6 months
* Cardiac surgery or percutaneous revascularization, MI, unstable angina, or CVA within the previous 30 days
* Antiarrhythmic drug therapy other than a beta-blocker within the previous 6 months
* Previous episode of sustained VT/VF or cardiac arrest, except in the setting of acute myocardial infarction or other reversible cause
* Life expectancy of less than one year from any non-cardiac cause
* Expected cardiac transplantation within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at high risk of arrhythmic event who do not have an ICD
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Reynolds, MD, Principal Investigator — VA Boston Healthcare System
Locations (19):
- United States (19):
  - VA GLAHS - David Geffen School of Medicine at UCLA, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Cardiovascular Consultants Medical Group, San Ramon, California
  - Cardiovascular Consultants Medical Group, Walnut Creek, California
  - St Francis Hospital and Medical Center, Hoffman Heart Institute, Hartford, Connecticut
  - Jim Moran Heart & Vascular Center, Fort Lauderdale, Florida
  - Florida Institute for Cardiovascular Care, Hollywood, Florida
  - Cardiac Disease Specialists, Atlanta, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - VA Boston Healthcare System, West Roxbury, Massachusetts
  - Michigan Heart, PC, Ypsilanti, Michigan
  - Mid America Heart Institute / Saint Luke's Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - St. Michael's Medical Center, Newark, New Jersey
  - Good Samaritan Hospital, Dayton, Ohio
  - Heart Institute of the Cascades, Bend, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina